CLINICAL TRIAL: NCT05810259
Title: Assessing the Effectiveness of Digital Wellness Modules on Perceived Quality of Life Via a Randomized Control Trial
Brief Title: Assessing the Effectiveness of Digital Wellness Modules on Perceived Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Caravan Wellness (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000034914; 000 (Other: CTGTY)
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Wellness; Quality of Life; Anxiety; Depression
Keywords: digital wellness interventions; wellness; mental health; mindfulness; exercise
MeSH Terms: conditions — Anxiety Disorders; Depression; Psychological Well-Being; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Mindfulness (Experimental): Participants will take part in 7 repeating digital mindfulness modules using the Caravan Wellness App.
  Interventions: Device: Caravan Wellness app
- Light to Moderate Physical Activity (Experimental): Participants will take part in 7 repeating light to moderate physical activity digital wellness modules using the Caravan Wellness App.
  Interventions: Device: Caravan Wellness app
- Control (No Intervention): A no intervention group that will not be using the Caravan Wellness App.

INTERVENTIONS:
Device: Caravan Wellness app — Caravan Wellness is a digital platform that offers brief mindfulness and light to moderate physical activity modules, among many others (e.g., Pilates, Yoga, Barre, meditation, etc.), to enhance overall individual well-being.
  Arms: Light to Moderate Physical Activity; Mindfulness

SUMMARY:
The study will examine the role of digital wellness modules (brief mindfulness and light to moderate physical exercise) delivered through a smartphone wellness application and their short-term effects on health behavior motivation and change, and longer-term quality of life and non-pathological affective states.

DETAILED DESCRIPTION:
Primary Objective: The primary objective of this parallel-assignment longitudinal study is to determine whether the digital wellness modules (e.g., mindfulness and light to moderate physical activity) increase quality of life and decrease stress, anxiety, and depression, as mediated by health behavior motivation and change in a healthy population of adults. Secondary Objective(s): The secondary objective is to ascertain qualitatively through deductive thematic analysis specific themes of a) key drivers of health behavior change; b) types of motivations that drive health behavior change, and c) implementation of sustained health behavior change.

The study will be conducted virtually by Yale University researchers.

ELIGIBILITY:
Inclusion Criteria:

* Resides in United States

Exclusion Criteria:

* Any individual who endorses any of the following criteria will be excluded from participation in this study:
* Positive Health Screening Questions, as measured by the Health Screening Questionnaire (HSQ):

  * Pain, discomfort or pressure in the chest, difficulty breathing or shortness of breath, dizziness, fainting, or blackout, blood pressure with systolic greater than 140 or diastolic greater than 90, diagnosed or treated for any heart disease, heart murmur, chest pain (angina), palpitations (irregular beat), or heart attack, heart surgery, angioplasty, or a pacemaker, valve replacement, or heart transplant, resting pulse greater than 100 beats per minute, any arthritis, back trouble, hip /knee/joint /pain, or any other bone or joint condition, personal experience or doctor's advice of any other medical or physical reason that would prohibit the participant from doing light to moderate physical exercise, personal physician's recommendation against participating in light to moderate physical exercise because of asthma, diabetes, epilepsy or elevated cholesterol or a hernia.
* Positive Psychiatric Disorders Screening Questions:

  * Positive screen for depression, excluding suicide (PHQ-8) cutoff score > 6
  * Positive screen for panic (SMPD) cutoff score > 2
  * Positive screen for generalized anxiety (GAD-7) cutoff score > 10
  * Positive screen psychosis (PDSQ) via psychosis section, cutoff score > 3
  * Positive screen mania via the Altman Self-Rating Mania Scale (ASRM) cutoff score > 6

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Mindfulness assessed by the Five Facet Mindfulness Questionnaire (FFMQ) | baseline, 1 Month follow up, 3 Month follow up
  The FFMQ is a 39-item questionnaire created to further explore the facet structure of mindfulness in daily life as a construct. It is composed of five component skills which contribute to mindfulness, non-reactivity to inner experiences (7 items), observing (8 items), acting with awareness (8 items), non-judging of inner experiences (8 items), and describing (8 items). Items are rated on a 5-point Likert- type scale, ranging from 1 (never or very rarely true) to 5 (very often or always true). Higher scores indicate more mindfulness.
Change in Exercise Behavior assessed by the Behavior Regulation Exercise Questionnaire, Third Version (BREQ-3) | baseline, 1 Month follow up, 3 Month follow up
  The BREQ-3 is a 24-item scale with five factors that measure external, introjected, identified, and intrinsic forms of regulation of exercise behavior based on Deci & Ryan's continuum conception of extrinsic and intrinsic motivation, described by organismic integration theory. Each item is scored on a five-point Likert scale, ranging from 0 ("Strongly Disagree") to 4 ("Strongly Agree"). Higher scores indicate an increase in exercise.
Utility of the Modules assessed by self report | up to Day 22
  Perceived utility of the modules will be assessed by self report using a one-item 5-point Likert scale = 0 (strongly disagree), 1 (disagree), 2 (agree), 3 (strongly agree), or 4 (undecided).
Daily stressors assessed using the Brief Daily Stressors Screening Tool (BDSST) | up to Day 22
  Daily stressors will be assessed using the BDSST, a short instrument for the recording of perceived general daily stressors in eight different areas of life. It is particularly suitable for use in large-scale studies or as a screening instrument for localizing areas of life where stress is particularly prevalent. A five-point Likert scale is used to measure the extent of the perceived stress experience from 0 ("Not at all") to 4 ("Very much") The higher the score, the more pronounced the subjective experience of general everyday stress.
Average number of minutes spent on Intervention | up to Day 22
  The average number of minutes per day spent on Intervention, as measured by self-report.
Change in health behavior motivation assessed using the Health Behavior Motivation Scale (HBMS) | baseline, 1 Month follow up, 3 Month follow up
  Change in health behavior motivation will be measured using the HBMS, a 30-item, five-point Likert scale that has a five-dimensional structure (i.e., intrinsic regulation, integrated and identified regulation, introjected regulation, external regulation, and amotivation). Scale ranges from 1 ("Definitely disagree") to 5 ("Definitely agree"). Higher scores indicate more health behavior motivation.
CHange in health behavior assessed using he Health Behavior Inventory-20 (HBI-20). | baseline, 1 Month follow up, 3 Month follow up
  Health behavior change will be measured using the HBI-20. The measure consists of a 20-items that factor into five subscales. Three subscales reflect health-promoting behaviors: Diet (five items), Preventive Care (seven items), and Medical Compliance (two items), and two subscales reflect health risk behaviors: Anger and Stress (three items), and Substance Use (three items). The health risk items are reverse-scored so that high scores on all subscales indicate a greater degree of health promotion and risk avoidance. Respondents are asked to rate the extent to which each item was self-descriptive, using a 7-point scale (e.g., 1 = always through 7 =never). Subscale scores are obtained by summing participants' responses (after reverse coding the risk items) and dividing them by the number of items.
Quality of life assessed using the Quality of Life Inventory (QOLI) | baseline, 1 Month follow up, 3 Month follow up
  The QOLI has 16 well-defined domains: health, self-esteem, goals and values, money, work, play, learning, creativity, helping, love, friends, children, relatives, home, neighborhood, and community. Within each domain, respondents are asked to rate the importance of that domain to their happiness on a 3-point scale: 0 = Not important, 1 = Important, and 2 = Extremely important. They then rate their satisfaction with each domain from -3 = Extremely, -2 = Somewhat, and -1 = A little dissatisfied to +1 = A little, +2 = Somewhat, and +3 = Extremely satisfied for each domain. The QOLI is scored by multiplying importance scores by satisfaction scores for each of the 16 domains, and then calculating an average across domains.
Change in stress and non-pathological anxiety and depression assessed using the Depression, Anxiety, and Stress Scale (DASS-21) | baseline, 1 Month follow up, 3 Month follow up
  The DASS-21 assesses key symptoms of depression, anxiety, and stress.The 21 items on the questionnaire comprise a set of three scales designed to assess depression, anxiety, and stress. The seven elements on each scale are rated on a Likert scale from 0 to 3 (0: "Did not apply to me at all," 1: "Applied to me to some degree or some of the time," 2: "Applied to me to a considerable degree or a good part of the time," and 3: "Applied to me very much or most of the time"). Scale scores are measured by summarizing the scores of the related items and then multiplying them by 2 to calculate the final score. Resulting ratings are then classified as: Depression: normal (0-4), mild (5-6), moderate (7-10), severe (11-13), or extremely severe (14+); Anxiety: normal (0-3), mild (4-5), moderate (6-7), severe (8-9), extremely severe (10+); Stress: normal (0-7), mild (8-9), moderate (10-12), severe (13-16), extremely severe (17+).

SECONDARY OUTCOMES:
Sleep quality assessed using the Pittsburgh Sleep Quality Index (PSQI) | baseline, 1 Month follow up, 3 Month follow up
  The PSQI is designed to evaluate overall sleep quality in clinical and non-clinical populations. The measure includes 19 self-reported items belonging to one of seven subcategories, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The questionnaire consists of a combination of Likert- type and openended questions (later converted to scaled scores using provided guidelines). Respondents are asked to indicate how frequently they have experienced certain sleep difficulties over the past month and to rate their overall sleep quality. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
Physical activity assessed using the International Physical Activity Questionnaire, Long Form (IPAQ-LF). | up to Day 22
  The IPAQ-LF is a 27-item survey that assesses the types of intensity of physical activity and sitting time. The scale asks respondents to rate during the last seven days engagement with physical activities.

CONTACTS AND LOCATIONS:
Overall Officials: David Klemanski, Psy.D., MPH, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No